CLINICAL TRIAL: NCT07184788
Title: Glofitamab，Polatuzumab Vedotin and GemOx in Refractory/Relapsed Aggressive B-Cell Lymphoma
Brief Title: G-Pola-GemOx in Refractory/Relapsed Aggressive B-Cell Lymphoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Navy General Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Liren Qian, Associate Chief Physician, Associate Professor, Navy General Hospital, Beijing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G-POLARGO
Record Dates: First submitted 2025-09-14; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Aggressive B-Cell Lymphoma
MeSH Terms: interventions — glofitamab; polatuzumab vedotin; Gemcitabine; Oxaliplatin; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Induction Therapy (Experimental): Patients were treated by G-Pola-GemOx as Induction Therapy
  Interventions: Drug: Glofitamab, Polatuzumab Vedotin, Gemcitabine, and Oxaliplatin as Induction Therapy

INTERVENTIONS:
Drug: Glofitamab, Polatuzumab Vedotin, Gemcitabine, and Oxaliplatin as Induction Therapy — Patients were treated by Glofitama(Cycle 1: D8, 2.5mg, D15, 10mg; followed by the target dose of 30mg on D1 of Cycle 2-12), Polatuzumab Vedotin(1.8mg/kg iv qd d1), Gemcitabine (1000 mg/m2 iv qd d2), Oxaliplatin (100 mg/m2 iv qd d2) as induction therapy.
  Other Names: G-Pola-GemOx

SUMMARY:
The goal of this phase 2 trial is to test the safety and efficacy of G-Pola-GemOx as induction therapy in patients with Refractory/Relapsed Aggressive B-Cell Lymphoma.

DETAILED DESCRIPTION:
The investigators will evaluate safety and efficacy of G-Pola-GemOx as induction therapy in Refractory/Relapsed Aggressive B-Cell Lymphoma. ORR(Overall response rate, progression-free survival (PFS), overall survival (OS), adverse events (AEs) will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed Aggressive B-Cell Lymphoma (Including but not limited to diffuse large B-cell lymphoma, mantle cell lymphoma, Burkitt lymphoma, high-grade B-cell lymphoma, etc. according World Health Organization (WHO) classification;
* Patient is ≥ 18 years of age at the time of signing the informed consent form (ICF).
* Patient must understand and voluntarily sign an ICF prior to any study-specific assessments/procedures being conducted;
* Patient is willing and able to adhere to the study visit schedule and other protocol requirements;
* Patient has not received chemotherapy previously.
* Anticipated life expectancy at least 3 months

Exclusion Criteria:

* Active or uncontrolled infections requiring systemic treatment within 14 days before enrollment.
* Any instability of systemic disease, including but not limited to severe cardiac, liver, kidney, or metabolic disease need therapy.
* Pregnant or lactating women

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2030-10-01 (Estimated); Study Completion 2031-10-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 1 year
  ORR was defined as the proportion of patients who achieved CR or PR as their best response

SECONDARY OUTCOMES:
Overall Survival (OS) | through study completion, an average of 2 years
  OS was defined as time from diagnosis to death from any cause or the last follow-up
Progression Free Survival (PFS) | 2 years]
  For patients in morphologic remission, documented relapse was considered progression. Relapse following complete remission(CR) is defined as reappearance of leukemic blasts in the peripheral blood or the finding of more than 5% blasts in the BM, not attributable to another cause (eg, BM regeneration after consolidation therapy) or extramedullary relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Liren Qian, Principal Investigator — Navy General Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No